CLINICAL TRIAL: NCT02153008
Title: Sofia Strep A FIA Field Study
Brief Title: Strep A FIA Field Study, Sofia
Status: Completed | Type: Observational
Sponsor: Quidel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-0142-07
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Group A Streptococcus
Keywords: Strep throat

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Symptomatic population for GAS: This study is a diagnostic study to aid in the detection of Strep throat. No intervention or medication is a part of this study.

SUMMARY:
To demonstrate the clinical performance of the Strep A FIA and Sofia, using throat swabs collected from symptomatic subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female, 3 years of age or older
2. Must currently be exhibiting one or more of the symptoms characteristic of pharyngitis to be eligible for inclusion in this study.

For example:

1. Acute onset of sore throat
2. Redness of the posterior pharyngeal wall
3. Difficulty/pain on swallowing
4. Fever, > 37.8º C (100ºF) at presentation or within past 24 hours
5. Pharyngeal exudate
6. Tender cervical lymphadenopathy
7. Absence of cough, runny nose or other upper respiratory symptoms.*
8. Other, symptoms specific to Strep A not listed above.

   * Must include at least one additional symptom from a-f and cannot be the only criteria used to meet inclusion for enrollment in the study.

Exclusion Criteria:

1. Subjects currently under treatment with antibiotics are not to be included in this study.
2. At clinical sites requiring informed consent, unable to understand and consent to participation; for minors this includes parent or legal guardian.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from the general population as they present to the clinical facility. Subjects must be exhibiting symptoms characteristic of pharyngitis, possibly GAS.
Sampling Method: Non-Probability Sample
Enrollment: 1708 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Detection of Group A Streptococcus | Within 5 minutes
  A throat swab specimen will be obtained and tested for the presence of Group A Streptococcus via the Sofia Analyzer

CONTACTS AND LOCATIONS:
Overall Officials: John D. Tamerius, PhD, Study Director — Quidel Corporation
Locations (7):
- United States (7):
  - Best Medical Group, LLC, Phoenix, Arizona
  - Gentle Medical Associates, Boynton Beach, Florida
  - Pediatrics by the Sea, Delray Beach, Florida
  - Teena Hughes, MD, Tampa, Florida
  - Twelve Corners Pediatrics, Rochester, New York
  - Veritas, PA, Belton, Texas
  - Advanced Pediatrics, Vienna, Virginia